CLINICAL TRIAL: NCT02843880
Title: Predictive Factors of Cytomegalovirus Reactivation or Cytomegalovirus Disease by Immunological Study of Immunocompetent Patients Hospitalized for Septic Shock
Brief Title: Prediction of Cytomegalovirus (CMV) Reactivation in Intensive Care Unit (ICU) by Immunological Study
Acronym: CMV-Réa
Status: Terminated | Type: Observational
Why Stopped: Problematic has become outdated in relation with current litterature advances.
Sponsor: AdministrateurDRC (Other)
Responsible Party: Sponsor-Investigator, AdministrateurDRC, Dr Maxime Lugosi, University Hospital, Grenoble
Organization: University Hospital, Grenoble (Other)
Other Study IDs: 2012/130
Record Dates: First submitted 2016-03-23; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: CMV Infection
Keywords: CMV reactivation; CMV disease; Predictive factors; Critically ill patients; Septic shock
MeSH Terms: conditions — Cytomegalovirus Infections; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Septic shock patients: Septic shock patients staying over 3 days mechanically ventilated in the ICU

SUMMARY:
Cytomegalovirus is a herpesviridae whose prevalence in general population is between 50 to 80%. In immunocompetent individuals, CMV remains latent in a number of cells, without any pathological consequence. Immunosuppression may reactivate the virus causing either a CMV-active infection or a CMV disease with attributable symptoms.

In Intensive Care Unit (ICU), 6 to 30 % of critically ill patients without classical immunosuppression, as those suffering from septic shock, present CMV reactivation. Our aim is to study the risk factors for developing viremia or CMV disease in ICU patients in septic shock without previous immunodepression and determine the relationship between viral reactivation and this acquired immunity alteration.

DETAILED DESCRIPTION:
Immunosuppression statuses causing both CMV active infection or disease are mainly consecutive to HIV infection, bone marrow or solid organ transplantation. However, in severely ill patients, as in septic shock, it has been proved that after a hyper-inflammatory phase occurred a negative control of the immunity, resulting in a paralysed or impaired immune system. The length and extent of this immunodeficiency is correlated with the duration of ICU stay, the occurrence of nosocomial infection and mortality.

A better understanding of CMV's natural history reactivation in the critically ill patient would better define the benefits from a specific therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* ICU admission for more than 3 days
* Admission for septic shock
* Patient with mechanical invasive ventilation

Exclusion Criteria:

* Immunodepression status before ICU admission (chemotherapy, bone marrow or solid organ transplantation, long time corticosteroid treatment, immunosuppressant therapy, HIV infection)
* Seronegative patient for CMV
* Patient under anti-virus treatment
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in ICU for septic shock, without previous immunodepression, and who will stay in ICU for over 3 days, mechanically ventialted
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of CMV disease | From Day 3 of ICU admission to the end of their stay in ICU (in average, from 6 days to 4 weeks)
  CMV disease is defined by occurence of viremia and/or an organ failure

SECONDARY OUTCOMES:
Mortality | Day 28
Length of ICU stay | About 90 days
Duration of mechanical ventilation | About 90 days
Occurence of nosocomial infections | About 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Universitary Hospital - Medical Intensive Care Station, Grenoble, France